CLINICAL TRIAL: NCT06711289
Title: Prediction of Hypotension After Spinal Anesthesia by Doppler Measurement of the Corrected Carotid Flow Time and the Peak Velocity Variation Within the Common Carotid Artery
Brief Title: Predicting If the Blood Pressure Will Drop After Spinal Anesthesia Using Ultrasound of the Neck
Status: Completed | Type: Observational
Sponsor: Catharina Ziekenhuis Eindhoven (Other)
Responsible Party: Principal Investigator, Joris Van Houte, Principal investigator, Catharina Ziekenhuis Eindhoven
Other Study IDs: W22.234
Record Dates: First submitted 2024-11-26; First posted 2024-12-02 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Spinal Anesthesia-induced Hypotension
Keywords: Spinal anesthesia-induced hypotension; Carotid Doppler ultrasound; Common carotid artery; Corrected carotid flow time; Peak velocity variation
MeSH Terms: interventions — Vital Signs; Anesthesia, Spinal

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Hypotensive patients: Patients who developed hypotension after the induction of spinal anesthesia.
  Interventions: Diagnostic Test: Carotid ultrasound measurement; Diagnostic Test: Vital sign measurement; Drug: Spinal anesthesia
- Normotensive patients: Patients who did not develop hypotension after the induction of spinal anesthesia.
  Interventions: Diagnostic Test: Carotid ultrasound measurement; Diagnostic Test: Vital sign measurement; Drug: Spinal anesthesia

INTERVENTIONS:
Diagnostic Test: Carotid ultrasound measurement — Pulsed-wave Doppler acquisition of the carotid artery. One acquisition will be made with the slow-speed setting (33 mm/s) and one with the medium-speed setting (66 mm/s).
Diagnostic Test: Vital sign measurement — Measurement of noninvasive blood pressure, at different time points before and after the induction of spinal anesthesia.
Drug: Spinal anesthesia — Following the standard of care, the patients received spinal anesthesia. The type and dosage of the local anesthetic were at the discretion of the treating anesthesiologist.

SUMMARY:
After a spinal injection, blood pressure might drop for a short time, similar to what happens with general anesthesia. This drop can be different for each person. An anesthesiologist will use medicine to bring the blood pressure back to normal. If this drop could be predicted in advance, it would help the anesthesiologist treat it faster, making the procedure even safer and preventing side effects like dizziness or nausea.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients of either sex who are scheduled for elective surgery under spinal anesthesia,
* Who fasted for 6 hours or more

Exclusion Criteria:

* Age <18 years old
* No informed consent for study participation
* Contra-indication for spinal anesthesia
* Emergency surgery
* Known poor left or right ventricular function / heart failure
* Moderate to severe valvular disease
* Atrial fibrillation
* Pacemaker rhythm
* Carotid artery stenosis > 50%
* History of cerebrovascular accident (CVA) or transient ischemic attack (TIA)
* History of cerebral trauma
* Pregnancy
* Neck complaints
* Morbid obesity (BMI > 40 kg/m2)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients scheduled for elective surgery under spinal anesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2023-04-12 (Actual); Primary Completion 2023-09-29 (Actual); Study Completion 2023-09-29 (Actual)

PRIMARY OUTCOMES:
Determine the predictive value of pre-anesthetic carotid parameters to predict spinal anesthesia-induced hypotension. | Prior to surgery.
  To determine the predictive value of pre-anesthetic corrected carotid flow time (ccFT) and peak velocity variation values for hypotension after induction of spinal anesthesia.

SECONDARY OUTCOMES:
Correlation between carotid parameters and blood pressure. | Trough study completion, an average of 30 minutes.
  To determine the correlation between the pre-anesthetic corrected carotid flow time (ccFT) and peak velocity variation on one hand and the maximal changes in systolic and mean arterial blood pressure after spinal anesthesia on the other hand.

OTHER OUTCOMES:
Intra-observer and inter-observer reproducibility of carotid Doppler parameters. | Prior to surgery.
  To determine the intra-observer and inter-observer reproducibility of Doppler parameters derived by two experienced sonographers.

CONTACTS AND LOCATIONS:
Overall Officials: Arthur Bouwman, Professor, Study Director — Catharina Ziekenhuis
Locations (1):
- Catharina Ziekenhuis, Eindhoven, North Brabant, Netherlands

IPD SHARING:
Plan to Share IPD: No
Patients did not give consent that their data would be used in studies other than spinal anesthesia-induced hypotension prediction.

REFERENCES:
- [Background] J. van Houte. The corrected carotid artery flow time and carotid peak velocity variation do not predict spinal anesthesia-induced hypotension: A prospective observational study. JCA Advances. 2024; 1: 1-8.
- [Derived] de Boer EC, van Houte J, Fernandes CD, Bakkes T, Muehlsteff J, Bouwman RA, Mischi M. Exploring the predictive value of carotid Doppler ultrasound and clinical features for spinal anesthesia-induced hypotension: a prospective observational study. Perioper Med (Lond). 2025 Mar 8;14(1):26. doi: 10.1186/s13741-025-00508-w. PMID 40057795